CLINICAL TRIAL: NCT07310329
Title: Effects of High-Dose Vitamin D Supplementation and Physical Exercise on Vitamin D Metabolites in Professional Football Players: A Pilot Study
Brief Title: High-Dose Vitamin D Supplementation and Exercise Effects on Vitamin D Metabolites in Professional Football Players
Acronym: VitD-Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Anna Książek, Associate Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AWF-VitD-Football-2024
Record Dates: First submitted 2025-11-27; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Vitamin D Deficiency (10 ng/mL to 30 ng/mL); Athletes; Football Players; Exercise Physiology
Keywords: 24,25-(OH)2D3; 3-epi-25-(OH)D3; dietary supplement; physical performance; athletes
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: a supplementation group receiving a single oral dose of 500,000 IU vitamin D₃ or a placebo group receiving identical placebo oil.
Who Masked: Participant
Masking Description: Single-blind design: participants were unaware of whether they received vitamin D₃ or placebo; the investigator administering supplements was unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation Group (SGP) (Experimental): Participants in this group received a single oral dose of 500,000 IU of vitamin D₃ (Vigantol Oil, P&G Health, Germany) 48 hours before the intra-squad football match (ISG). Blood samples were collected before supplementation and both before and after the ISG to evaluate changes in vitamin D metabolites.
  Interventions: Dietary Supplement: Vitamin D₃
- Placebo Group (PGP) (Placebo Comparator): Participants in this group received a single oral dose of placebo oil identical in color and consistency to the vitamin D₃ solution. Blood samples were collected at the same time points as in the supplementation group to assess vitamin D metabolite changes.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D₃ — A single oral dose of 500,000 IU vitamin D₃ (Vigantol Oil, P&G Health, Germany) was administered 48 hours before the intra-squad football match to assess its acute effects on vitamin D metabolite concentrations.
  Arms: Supplementation Group (SGP)
Other: Placebo — A single oral dose of vegetable oil matching the vitamin D₃ solution in color and consistency was administered 48 hours before the intra-squad football match.
  Arms: Placebo Group (PGP)

SUMMARY:
This randomized, single-blind, placebo-controlled pilot study investigated the effects of high-dose vitamin D₃ supplementation and football-specific physical exercise on vitamin D metabolite concentrations in professional male football players. The study aimed to evaluate the acute response of circulating vitamin D metabolites, including 25-(OH)D₃, 24,25-(OH)₂D₃, and 3-epi-25-(OH)D₃, following a single oral dose of 500,000 IU cholecalciferol combined with high-intensity intermittent exercise typical of competitive football.

Twenty professional football players from a Polish top-division club participated in the study. Participants were randomly assigned to either the supplementation group (SGP) receiving 500,000 IU of vitamin D₃ or the placebo group (PGP) receiving an identical volume of placebo oil. The intervention was administered 48 hours prior to an intra-squad game. Blood samples were collected at three time points: baseline (T3), pre-match (T4), and post-match (T5). The primary outcome was the change in serum 25-(OH)D₃ concentration. Secondary outcomes included changes in 24,25-(OH)₂D₃ and 3-epi-25-(OH)D₃ levels, as well as their ratios. The study also assessed whether physical exercise modulates vitamin D metabolism.

The findings demonstrated that high-dose vitamin D₃ supplementation significantly increased serum 25-(OH)D₃ (↑198%) and 3-epi-25-(OH)D₃ (↑444%) levels, while football-specific exercise itself induced moderate increases in vitamin D metabolites. The results suggest that skeletal muscle may play a key role in vitamin D storage and release in response to exercise. The supplementation was well tolerated, with no adverse events observed.

DETAILED DESCRIPTION:
This pilot study was designed to explore the combined effects of high-dose vitamin D₃ supplementation and acute physical exercise on vitamin D metabolism in professional football players. The study responds to growing scientific interest in understanding how vitamin D status influences performance, recovery, and muscle function in athletes. While most previous studies have focused on chronic, low-to-moderate supplementation, this trial examined the response to a single, pharmacological dose of cholecalciferol in a controlled experimental setting.

Study Design

The study employed a randomized, single-blind, placebo-controlled, parallel-group design. Participants were randomly assigned to one of two groups:

Supplementation Group (SGP) - received a single oral dose of 500,000 IU vitamin D₃ (Vigantol Oil, P&G Health, Germany);

Placebo Group (PGP) - received an identical amount of placebo (vegetable oil).

The supplementation was administered 48 hours before a standardized intra-squad football match (ISG), conducted under conditions simulating a competitive game. All players followed the same training schedule and diet during the study.

Participants

A total of 20 professional male football players (aged 18-35) from a Polish top-league club volunteered to participate. Inclusion criteria included active professional status, regular training participation, and no use of vitamin D or calcium supplements in the previous 3 months. Exclusion criteria included musculoskeletal injuries, metabolic disorders, or refusal to sign informed consent.

Measurements

Blood samples were collected at three time points:

T3: baseline (before supplementation),

T4: 48 hours post-supplementation (pre-match),

T5: immediately after the intra-squad game.

Serum concentrations of 25-(OH)D₃, 24,25-(OH)₂D₃, and 3-epi-25-(OH)D₃ were determined using LC-MS/MS. Additional biochemical variables (hemoglobin, glucose, testosterone, cortisol, ferritin, calcium, CK) were analyzed to monitor physiological status.

Outcomes

Primary Outcome: Changes in serum 25-(OH)D₃ concentrations after supplementation and exercise.

Secondary Outcomes: Changes in 24,25-(OH)₂D₃ and 3-epi-25-(OH)D₃ levels, metabolite ratios.

Ethics

The study was approved by the Ethics Committee of the Wroclaw University of Health and Sport Sciences (Resolution No. 1/2024, March 1, 2024). All participants signed written informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Male professional football players aged 18-35 years
2. Actively training and competing in the Polish first football league
3. No vitamin D or calcium supplementation during the previous 3 months
4. No injuries or illnesses affecting participation

Exclusion Criteria:

1. Current musculoskeletal injury or illness
2. Chronic metabolic, endocrine, or renal disorders
3. Use of vitamin D or calcium supplements
4. Refusal or inability to sign informed consent

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Changes in serum 25(OH)D₃ concentration | Baseline (before supplementation), 48 hours after supplementation, and immediately after the football match (2 days after supplementation).
  Serum concentrations of 25(OH)D₃ will be measured using isotope-dilution liquid chromatography-tandem mass spectrometry (ID-LC-MS/MS). The primary outcome assesses the effect of a single high-dose vitamin D₃ supplementation combined with physical exercise on 25(OH)D₃ concentration in professional football players.
Changes in serum 24,25-dihydroxyvitamin D₃ [24,25(OH)₂D₃] concentration | Baseline (T3), 48 hours post-supplementation (T4), and post-exercise (T5)
  To evaluate the effect of vitamin D₃ supplementation and physical exercise on 24,25(OH)₂D₃ levels using ID-LC-MS/MS.

SECONDARY OUTCOMES:
Changes in metabolite ratios (25(OH)D₃:24,25(OH)₂D₃ and 25(OH)D₃:3-epi-25(OH)D₃) | Baseline (before supplementation), 48 hours after supplementation, and immediately after the football match (2 days after supplementation).
  To assess changes in the ratios between major vitamin D metabolites as indicators of metabolic transformation rate and vitamin D turnover in response to supplementation and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Książek, PhD Eng.; Associate Professor, Principal Investigator — Department of Biological Principles of Physical Activity ; Wroclaw University of Health and Sport Sciences
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Dolnyśląsk, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy considerations and the specific nature of the study population (professional athletes). Aggregated data are available upon reasonable request to the corresponding author.

REFERENCES:
- [Result] Mieszkowski J, Stankiewicz B, Kochanowicz A, Niespodzinski B, Kowalik T, Zmijewski M, Kowalski K, Rola R, Bienkowski T, Antosiewicz J. Ultra-Marathon-Induced Increase in Serum Levels of Vitamin D Metabolites: A Double-Blind Randomized Controlled Trial. Nutrients. 2020 Nov 25;12(12):3629. doi: 10.3390/nu12123629. PMID 33255807